CLINICAL TRIAL: NCT02582606
Title: Effects of the Constancy of Daily Meal Pattern on Energy Balance, Glucose Profiles and Plasma Lipoproteins in Obese Women
Brief Title: Meal Pattern and Metabolic Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Elizabeth Simpson, Senior Research Fellow, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: P3/15
Record Dates: First submitted 2015-10-16; First posted 2015-10-21 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Insulin Resistance
Keywords: Insulin Resistance; Meal pattern; Obese
MeSH Terms: conditions — Insulin Resistance; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regular (Experimental): Regular meal pattern
  Interventions: Other: Regular meal pattern
- Irregular (Experimental): Irregular meal pattern
  Interventions: Other: Irregular meal pattern

INTERVENTIONS:
Other: Regular meal pattern — a 14-day period of eating 6 meal per day
  Arms: Regular
Other: Irregular meal pattern — a 14-day period of eating between 3 and 9 meal per day
  Arms: Irregular

SUMMARY:
In this study investigators will compare the health effect of two different meal patterns. In one, participants will consume food according to an 'irregular meal pattern' (minimum 3 meals, maximum 9 meals per day) and in the other 'regular meal pattern' (6 meals per day) for two weeks. The energy requirement of the participants will be calculated to maintain body weight during the study. Participants will be provided with all the food to be consumed during the study.

Initially, interested individuals will attend a screening visit in which they will complete questionnaires on medical health, eating habits and physical activity. Height, weight and waist circumference will be measured at this visit. Thereafter, participants will be assigned to a 2-week period following one of the two meal-patterns. There will be a 2-week period between the two interventions when they will consume their normal diet and at the end of this, participants will undertake the next meal pattern. During the two phases participants will be asked to wear an armband (which detects movement and measures heat loss), to assess their energy expenditure and an interstitial glucose monitoring device will be worn for seven days. Before and after each 2-week intervention, participants will come to the laboratory for a mixed-meal tolerance test. Blood samples will be obtained before and for 3hrs after eating to evaluate the health effects of the meal patterns. Energy expenditure will be measured by ventilated-hood indirect calorimetry and the armband device. At the end of the 3hr post prandial period, participants will be offered an ad libitum pasta lunch and be asked to eat until they feel comfortably full.

During each of the 2-week periods, participants will be asked to record their food intake and record their appetite sensations on specific days.

DETAILED DESCRIPTION:
Background. Greater variation in meal pattern from day to day might affect energy balance and, in consequence, the control of body weight. However, studies which have evaluated the impact of an irregular meal pattern on energy metabolism, in adults, are few. Several experimental studies by Farshchi et al. have shown that there are potentially important negative health consequences associated with erratic/irregular eating patterns. Higher fasting levels of total-cholesterol and low density lipoprotein (LDL)-cholesterol, a decrease in thermic effect of food (TEF), and reduced insulin sensitivity, were observed in healthy women after 14 days of irregular eating. Subsequent studies have confirmed this in overweight subjects and also provided evidence of alterations in subjective appetite which may influence ad-libitum food intake (Lara et al, unpublished).

Recently, experimenters have shown a decrease in thermogenesis in response to a test meal, and greater postprandial blood glucose concentration in 11 normal weight women following two-weeks of irregular eating in contrast to a regular pattern.

The present study will study the effect of an irregular meal pattern in obese women who demonstrate fasting insulin resistance (IR).

Aims:

to investigate the effects of meal pattern on energy expenditure, postprandial thermogenesis, postprandial blood glucose, fasting lipid profile and fasting insulin sensitivity in obese women with insulin resistance.

Experimental protocol. 10 women with a homeostatic model assessment - insulin resistance (HOMA-IR) ≥1.8, body mass index between 28 and 40 kg/m2, aged 18-45 years, and who are otherwise healthy, will be recruited. Interested individuals will have an initial medical screening to confirm suitability. Those who are recruited will be asked to then complete a 7 days food diary before participating in the study. The whole study will last for a total of 6 weeks. During the first 2 weeks participants will adopt one of two meal patterns, followed by a two-week washout period during which they resume their habitual diet and meal pattern. A second 2-week intervention will then follow, in which the alternative meal pattern is adopted. The meal patterns will be 1) regular - 6 daily meals or snacks for 2 weeks, or 2) irregular - a different number (between 3 and 9) of meals/snacks every day. Allocation of the order in which the diets are tested will be randomized at the point of recruitment with participant number assigned sequentially. All foods to be consumed during weeks1, 2, 5 and 6 will be provided free of charge, and will comprise foods commonly consumed in the British diet, in quantities designed to keep body weight constant during the study. Participants will complete food diaries over the whole study period. They will be asked to wear a 'SenseWear' armband (SWA) device (attached to an upper arm) to allow physical activity and energy expenditure to be estimated during weeks1, 2, 5 and 6. Participants will attend the laboratory on the 6th day of each intervention phase to have a continuous interstitial glucose monitoring probe inserted in the subcutaneous abdominal fat pad at the level of the umbilicus. Participants will measure their blood glucose four times a day, using a fingerprick sample and pocket glucose analyser, to calibrate the continuous glucose monitor. After three days participants will be asked to come back to have this device removed.

Subjective appetite (hunger, fullness, etc.) will be assessed using visual analogue scales (VAS) during the intervention (at the end of each week, and whilst the glucose monitor is being worn).

Before and after each intervention period, participants will visit the laboratory after fasting overnight. At 8:30 am a cannula will be inserted into a hand vein, with the hand placed in a hot-air box, for subsequent blood sampling. Indirect calorimetry will be performed to determine energy expenditure, carbohydrate and lipid oxidation rates and changes in the thermic response to a milkshake test drink providing 10 kcals/kg body weight, and comprising 35% of energy as fat, 15% as protein, and 50% as carbohydrate. The SWA device will also be placed on the upper left arm to estimate energy expenditure during the laboratory visit. Blood samples will be obtained before and every 15 minutes for 3 hours after eating. Indirect calorimetry and SWA will be measured concurrently for the duration of the laboratory visit. Fasting blood samples will be used to measure total-, high density lipoprotein (HDL)-, LDL-, and very low density lipoprotein (VLDL)-cholesterol, triglycerides, glucose and insulin. Blood samples obtained after the test drink will also be used to measure glucose, insulin and hormones related to appetite. After the 3hr postprandial period, a test meal (pasta) will be provided as ad-libitum meal and participants will be asked to fill VAS to assess subjective appetite sensations.

Measurable end points of the study

* 24hr Energy expenditure during the two phases (irregular versus regular meal pattern)
* Fasting lipids, insulin, glucose and glucose profiles during the continuous monitoring
* Insulin, glucose and gut hormone (Glucagon-Like Peptide 1, Ghrelin and Peptide YY) responses to the test drink
* Postprandial thermogenic response to a test drink
* Ratings of subjective appetite during the study Sample size and statistical power Using 1 sample t-test model, power calculated at the level of 0.8. Primary end point = difference in thermic effect of food 'TEF' (kcal/min) over 180min. Results obtained from study previous studies indicated the incremental area under the TEF curve after regular eating was 25.8 (SD 6.8) kcal and after irregular eating was 14.8 (SD 11.7) kcal. With a cross-over design, 10 subjects in each group would be able to detect a change in TEF with the power of 80% at the level of 0.05 significance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy;
* BMI 28 - 40 kg/m2
* Insulin resistance, HOMA ≥ 1.5
* Weight stable during the last 3 months (self-reported weight change < ± 2 kg)

Exclusion Criteria:

* history of serious disease as assessed by a medical screening questionnaire
* taking any medication except for the oral contraceptive pill.
* Smokers
* high alcohol consumers (< 2-3 units/day),
* pregnant/lactating
* irregular menstrual cycles
* dieting/seeking to lose weight
* clinical symptoms of depression (Beck)
* eating disorder (EAT-26)
* allergy or intolerance to any of the foods provided during each study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2014-02; Primary Completion 2014-10 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in fasting insulin sensitivity, as measured by HOMA-IR | 14 days
  insulin sensitivity assessed using fasting circulating insulin and glucose concentration and the HOMA-insulin resistance (IR) index

SECONDARY OUTCOMES:
Change in postprandial circulating insulin concentration | 14 days
  assessed during the mixed meal tolerance test using serum insulin concentration
Change in thermic effect of food | 14 days
  fasting and postprandial energy expenditure assessed by indirect calorimetry during laboratory visits
Change in subjective appetite | 14 days
  Will be assessed by Visual Analogue Scale during the intervention and throughout the mixed meal tolerance test.
Change in appetite hormones | 14 days
  Circulating level of leptin, adiponectin, glucagon-like peptide1, peptide YY and ghrelin before and during the mixed meal tolerance test.
Change in fasting cholesterol | 14 days
  will be assessed before each mixed meal tolerance test

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Macdonald, PhD, Principal Investigator — University of Nottingham
Locations (1):
- David Greenfield Human Physiology Unit, University of Nottingham Medical School, Nottingham, Notts, United Kingdom

REFERENCES:
- [Background] Farshchi HR, Taylor MA, Macdonald IA. Decreased thermic effect of food after an irregular compared with a regular meal pattern in healthy lean women. Int J Obes Relat Metab Disord. 2004 May;28(5):653-60. doi: 10.1038/sj.ijo.0802616. PMID 15085170
- [Background] Farshchi HR, Taylor MA, Macdonald IA. Regular meal frequency creates more appropriate insulin sensitivity and lipid profiles compared with irregular meal frequency in healthy lean women. Eur J Clin Nutr. 2004 Jul;58(7):1071-7. doi: 10.1038/sj.ejcn.1601935. PMID 15220950
- [Background] Farshchi HR, Taylor MA, Macdonald IA. Beneficial metabolic effects of regular meal frequency on dietary thermogenesis, insulin sensitivity, and fasting lipid profiles in healthy obese women. Am J Clin Nutr. 2005 Jan;81(1):16-24. doi: 10.1093/ajcn/81.1.16. PMID 15640455
- [Derived] Alhussain MH, Macdonald IA, Taylor MA. Impact of isoenergetic intake of irregular meal patterns on thermogenesis, glucose metabolism, and appetite: a randomized controlled trial. Am J Clin Nutr. 2022 Jan 11;115(1):284-297. doi: 10.1093/ajcn/nqab323. PMID 34555151